CLINICAL TRIAL: NCT07294859
Title: A Prospective Clinical Study on the Predictive Value of CEUS and Super-resolution Imaging Technology for Renal Function Outcome in Patients After Partial or Radical Nephrectomy
Brief Title: Contrast-enhanced Ultrasound and Super-resolution Imaging Predict Renal Function Outcome After Nephrectomy
Status: Recruiting | Type: Observational
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Le Qu, Associate chief urologist, Jinling Hospital, China
Other Study IDs: DZQH-KYLL-25-37
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Nephrectomy; Renal Cell Cancer; AKI - Acute Kidney Injury
MeSH Terms: conditions — Carcinoma, Renal Cell; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients scheduled for radical nephrectomy
- Patients scheduled for partial nephrectomy

SUMMARY:
The goal of this prospective cohort study is to evaluate the predictive value of Contrast-Enhanced Ultrasound (CEUS) and Super-Resolution Imaging (SRI) technologies regarding renal function outcomes in patients with renal cell carcinoma (RCC) undergoing partial or radical nephrectomy. The main questions it aims to answer are:

Can quantitative parameters of renal microcirculation and microvascular structure derived from CEUS and SRI predict long-term renal function (defined as New Baseline eGFR for radical nephrectomy and Recovery from Ischemia for partial nephrectomy)? Can these imaging parameters accurately predict the occurrence, severity, and early recovery of postoperative acute kidney injury (AKI)? Researchers will monitor the dynamic evolution of renal blood flow and microvascular density by comparing the affected kidney to the contralateral healthy kidney before and after surgery to see if these biomarkers correlate with clinical outcomes.

Participants will:

Undergo CEUS and SRI examinations before surgery and at specific time points after surgery (e.g., within 7 days) to visualize renal microvasculature.

Provide blood and urine samples for standard laboratory tests (such as serum creatinine and Cystatin C) to assess kidney function during hospitalization.

Attend follow-up visits at 1, 3, 6, 9, and 12 months post-surgery to monitor long-term renal recovery and complete necessary imaging assessments (CT or Ultrasound).

DETAILED DESCRIPTION:
This study is a prospective cohort study aimed at evaluating the predictive value of contrast-enhanced ultrasound and super-resolution imaging techniques for renal function outcomes in patients after nephrectomy. The study intends to include approximately 285 patients with renal cell carcinoma who are scheduled to undergo partial nephrectomy or radical nephrectomy. The core of this study is to non-invasive and quantitatively monitor the microcirculation perfusion (such as hemodynamic parameters) and microvascular structure (such as microvascular density and glomerular density) of the affected and healthy kidneys at multiple time points before and after the operation by applying contrast-enhanced ultrasound and super-resolution imaging techniques, and simultaneously collect clinical data.

The main contents of this study include: longitudinal observation of the dynamic evolution patterns of renal microcirculation parameters before and after the operation; Analyze the correlations between these imaging parameters and the occurrence, severity and prognosis of postoperative acute kidney injury, and simultaneously explore the association between the occurrence and development of early AKI and long-term renal function changes; Ultimately, the goal is to combine predictive imaging parameters with traditional clinical variables (such as age, preoperative renal function, etc.) to construct integrated mathematical models for different surgical methods (partial nephrectomy and radical nephrectomy), in order to accurately predict the early (postoperative acute kidney injury) and long-term renal function (such as new baseline estimated glomerular filtration rate) of patients. Meanwhile, considering the compensatory function of contralateral renal function after PN, Rec-Ischemia was adopted as the primary endpoint indicator to evaluate the changes of ipsilateral postoperative renal function in patients after PN. This study is expected to provide innovative imaging biomarkers and decision support for individualized management and early intervention of renal function after nephrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Fully understood and voluntarily signed the informed Consent Form (ICF);
* Age: > 18 (at the time of signing the informed consent form); Gender is not limited.
* Preoperative eGFR > 45ml/min/1.73m2 (corrected CKD-EPI formula);
* After the clinician formulates the treatment plan and communicates with the patient, they decide whether to perform radical nephrectomy or partial nephrectomy.
* ECOG score: 0-2 points;
* Be willing and able to abide by the visits, treatments, laboratory tests and other procedures of the research plan.

Exclusion Criteria:

* Patients with solitary kidney or severe contralateral renal insufficiency (eGFR < 15ml/min/1.73m2);
* Preoperative reliance on renal replacement therapy (such as dialysis, etc.);
* Those who fail to complete the nephrectomy as planned during the operation;
* Patients with lymph node metastasis, distant metastasis or venous tumor thrombus;
* The healthy kidney has undergone radiotherapy, ablation or other surgeries.
* Have a history of allergy to ultrasound contrast agents;
* Have any contraindications for contrast-enhanced ultrasound, such as right-to-left shunt, severe pulmonary hypertension, etc.
* Patients with hemodynamic instability, including those with persistent hypotension (blood pressure < 90/60 MMHG), uncontrollable heart failure, active bleeding (such as gastrointestinal and cerebral hemorrhage, etc.), or those with a bleeding tendency and hemoglobin < 60g/L and/or platelet count < 50×109/L;
* Accompanied by structural abnormalities of the urinary system or functional abnormalities that cannot be corrected in a short time (such as duplicate kidneys, polycystic kidneys, horseshoe kidneys, isolated kidneys, renal artery stenosis > 50%, urinary tract obstruction, and previous history of kidney surgery, etc.), long-term indwelling of urinary catheters, etc.
* There are other diseases that limit life expectancy to less than six months;
* Previous (≤30 days before randomization) or concurrent participation in another clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for radical or partial nephrectomy who met all inclusion criteria but did not meet any exclusion criteria
Sampling Method: Probability Sample
Enrollment: 285 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
new baseline estimates glomerular filtration rate(NB-eGFR) | 12 months after nephrectomy
  NB-eGFR is defined as multiple eGFR tests conducted within 3 to 12 months after surgery, and the last eGFR measurement value within this time window (the calculation of eGFR uses the corrected CKD-EPI formula)
Rec-Ischemia | 12 months after partial nephrectomy
  This outcome is mainly applicable to patients undergoing partial nephrectomy. It is defined as the ratio of the ipsilateral GFR retention rate to the renal parenchymal retention rate (PPVP), that is, the degree of functional recovery of the retained renal parenchyma per unit. The calculation formula is Rec-Ischemia= ipsilateral GFR retention rate /PPVP×100%13.
  Ipsilateral GFR retention rate = postoperative ipsilateral GFR/ preoperative ipsilateral GFR×100%, PPVP= postoperative ipsilateral renal parenchymal volume/preoperative ipsilateral renal parenchymal volume ×100%. The predicted ipsilateral GFR after surgery = the total postoperative GFR× the expected retained SRF of the affected kidney. The expected retained SRF of the affected kidney = the parenchymal volume of the affected kidney/(the parenchymal volume of the affected kidney + the parenchymal volume of the contralateral kidney).

CONTACTS AND LOCATIONS:
Locations (1):
- Jinling Hospital, Affiliated Hospital of Medical School, Nanjing University, Nanjing, Jiangsu, China